CLINICAL TRIAL: NCT01452945
Title: Prospective Observational Study Evaluating the Use of Bedside Lung Ultrasound in Young Children Presenting to the Emergency Department With Wheezing
Brief Title: Bedside Lung Ultrasound in Young Children Presenting to the Emergency Department (ED) With Wheezing
Status: Completed | Type: Observational
Sponsor: Children's National Research Institute (Other)
Responsible Party: Principal Investigator, Joanna Cohen, Assistant Professor of Pediatrics and Emergency Medicine, Children's National Research Institute
Other Study IDs: Pro00002000
Record Dates: First submitted 2011-10-13; First posted 2011-10-17 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2015-05

CONDITIONS: Wheezing; Bronchiolitis
MeSH Terms: conditions — Respiratory Sounds; Bronchiolitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Young children presenting to the Emergency Department (ED) with wheezing often have prolonged stays in the ED or even get admitted to the hospital. This is a prospective observational study in which the investigators will use bedside 2D ultrasound to evaluate the lung ultrasound findings in children less than 24 months presenting to the ED with wheezing.

The investigators hypothesize that children less than 24 months presenting to the Emergency Department with wheezing will have a range of lung ultrasound findings that will include normal findings, B lines, subpleural consolidations, and pleural effusions. The investigators also hypothesize that the findings will be reproducible between two equally trained providers.

The investigators also hypothesize that lung ultrasound findings patients 0-24 months presenting to the ED with wheezing will correlate with specific clinical outcomes. An exploratory analysis will be performed to look for correlations between lung US findings and acute severity, final diagnosis, presenting symptoms, prematurity, risk factors for atopy, response to treatment and radiologic or viral studies if performed.

DETAILED DESCRIPTION:
Specific Aim 1: To qualify lung US findings in a convenience sample of young children presenting to the ED with bronchiolitis with review by a second provider to determine the reproducibility of the findings.

reproducibility of the findings.

Hypothesis 1a: Children less than 24 months presenting to the Emergency Department with wheezing will have a range of lung ultrasound findings that will include normal findings, B lines, subpleural consolidations, and pleural effusions.

Hypothesis 1b: Findings will be reproducible between two equally trained providers.

Specific Aim 2: The frequency of B lines, subpleural consolidations, and pleural effusions on lung US in a convenience sample of patients 0-24 months presenting the ED with wheezing will be quantified using continuous variable means and standard deviations. An exploratory analysis will be performed to look for correlations between lung US findings and clinical outcomes including discharge from the ED or admission to the hospital, including the intensive care unit, and length of stay in the ED. A further exploratory analysis will be done to look for correlations between lung ultrasound findings and acute severity, final diagnosis, presenting symptoms, prematurity and risk factors for atopy.

Hypothesis 2a: The presence of B lines, subpleural consolidations, and pleural effusions on lung US in a convenience sample of patients 0-24 months presenting the ED with wheezing will correlate with specific clinical outcomes.

Hypothesis 2b: The presence of B lines, subpleural consolidations, and pleural effusions on lung US in a convenience sample of patients 0-24 months presenting the ED with wheezing will positively correlate with a history of prematurity and negatively correlate with a history consistent with atopy.

ELIGIBILITY:
Inclusion Criteria:

* Age less than or equal to 24 months
* Presenting to the pediatric ED with wheezing

Exclusion Criteria:

* On home oxygen at baseline
* Cyanotic congenital cardiac disease (including: ToF, TAPVR, HLHS, d-TGA, TA, pulm atresia, critical pulm stenosis, but not including VSD, ASD, Coarctation of the Aorta)
* Endotracheal tube or tracheostomy in place and/or receiving mechanical ventilation
* Transferred from an outside hospital

Max Age: 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children 0-24 months presenting to a pediatric Emergency Department with wheezing
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2012-10; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joanna S Cohen, MD, Principal Investigator — Children's National Research Institute
Locations (1):
- Children's National Medical Center Division of Emergency Medicine, Washington D.C., District of Columbia, United States

REFERENCES:
- [Background] Volpicelli G, Mussa A, Garofalo G, Cardinale L, Casoli G, Perotto F, Fava C, Frascisco M. Bedside lung ultrasound in the assessment of alveolar-interstitial syndrome. Am J Emerg Med. 2006 Oct;24(6):689-96. doi: 10.1016/j.ajem.2006.02.013. PMID 16984837
- [Background] Lichtenstein D, Meziere G, Biderman P, Gepner A, Barre O. The comet-tail artifact. An ultrasound sign of alveolar-interstitial syndrome. Am J Respir Crit Care Med. 1997 Nov;156(5):1640-6. doi: 10.1164/ajrccm.156.5.96-07096. PMID 9372688
- [Background] Copetti R, Cattarossi L, Macagno F, Violino M, Furlan R. Lung ultrasound in respiratory distress syndrome: a useful tool for early diagnosis. Neonatology. 2008;94(1):52-9. doi: 10.1159/000113059. Epub 2008 Jan 15. PMID 18196931
- [Background] Caiulo VA, Gargani L, Caiulo S, Fisicaro A, Moramarco F, Latini G, Picano E. Lung ultrasound in bronchiolitis: comparison with chest X-ray. Eur J Pediatr. 2011 Nov;170(11):1427-33. doi: 10.1007/s00431-011-1461-2. Epub 2011 Apr 6. PMID 21468639